CLINICAL TRIAL: NCT06464497
Title: Whole Foods for Teens: A Pilot Dietary Intervention to Reduce Body Adiposity in Adolescents With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nadia Markie Sneed, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 240866
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Childhood; Diet, Healthy; Body Weight Changes
MeSH Terms: conditions — Pediatric Obesity; Body Weight Changes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Foods Counseling Group (No Intervention): Participants randomized to the "usual care" group will receive a MyPlate Plan that follows a conventional Dietary Guidelines for Americans (DGA) diet which is considered a healthy diet pattern for adolescents with obesity. This diet intervention will encourage the consumption of a whole foods "dietary patterns" such as a wide variety of fruits, vegetables, proteins, seafood, dairy and whole grains. Physical activity will be encouraged per MyPlate guidelines and will be reported on the MyPlate plan daily. At the end of each week, study personnel and/or the study RDN will follow up with the participants to review the food checklists. At this time personnel will address diet-related questions and provide guidance on diet adherence.
- Whole Foods MyPlate Group (Experimental): Adolescents and adults randomized to the "intervention group" will receive a MyPlate Plan to support daily food group and macronutrient goals that align with the whole foods diet per caloric needs. The 8-week intervention will consist of rotating menus (per above) and bi-weekly groceries of mostly fruits and vegetables delivered to family's homes that align with the study menus to support adherence.
  Interventions: Behavioral: Whole Foods MyPlate Group

INTERVENTIONS:
Behavioral: Whole Foods MyPlate Group — Families will receive 4-weeks of rotating menus that have been designed as a part of our preliminary work and will be adapted to support adherence with the adolescent in mind (e.g., school lunch options, on-the-go snacks). Menus and diet recommendations will align with the current macronutrient nutritional goals outlined by the 2020-2025 DGA for age-sex groups. Participants will be encouraged to eat ad libitum (i.e., as desired until full) without calorie restrictions. MyPlate will be used by participants to implement the diet. During the study, adolescents and adults in the intervention group will receive a MyPlate Plan to support daily food group and macronutrient goals that align with the whole foods diet per caloric needs.
  Arms: Whole Foods MyPlate Group

SUMMARY:
This study will address the following aims:

Aim 1: Conduct an 8-week pilot RCT to examine the effects of a whole foods diet intervention on body adiposity in adolescents with obesity.

Aim 1a (Primary): Evaluate intervention effectiveness on total fat mass following the 8-week intervention.

Hypothesis 1a: Adolescents randomized to the whole foods intervention will have lower total fat mass (kg) at the 8-week follow-up than those in the control group.

Aim 1b: Evaluate intervention effectiveness on anthropometric changes following the 8-week intervention.

Hypothesis 1b: Adolescents randomized to the whole foods intervention will have lower weight, BMI-z scores and/or waist circumference at the 8-week follow-up than those in the control group.

Secondary Aims:

Aim 2: Conduct an 8-week pilot RCT to examine the effects of a whole foods diet intervention on diet quality in adolescent and parent pairs during the study period.

Hypothesis 2: Adolescents and parents randomized to the whole foods intervention will have higher diet quality scores at the 8-week follow-up than those in the control group.

Aim 3: Conduct post-intervention family focus groups to identify how individual/family needs and preferences and social determinants of health (SDOH) may be perceived barriers and/or facilitators of diet adherence to a whole foods diet pattern.

DETAILED DESCRIPTION:
For adolescents with obesity, a healthy diet pattern is recommended as a first-line non-pharmacological treatment. Yet, despite decades of research, there is inconclusive evidence from randomized clinical trials (RCT) to support an optimal dietary pattern to treat adolescent obesity. While observational data has linked poor-quality diet patterns high in calories, fat, and refined carbohydrates to greater body adiposity in adolescents, some research suggests that dietary patterns that emphasize high-quality whole foods (e.g. Mediterranean, low-glycemic load) not only improve diet quality but can also effectively reduce body adiposity and improve metabolic outcomes (e.g., insulin resistance) without the need for calorie restrictions. However, for adolescents with obesity, adherence to a healthy diet pattern requires the involvement of the whole family, with the potential to improve diet quality and reduce body adiposity and its associated metabolic complications. Unfortunately, weaknesses of past studies include 1) a failure to intervene upon diet quality at the family level to modify adolescent dietary behaviors, and 2) a lack of consideration for how individual/family needs and social determinants of health (SDOH) impact diet adoption. To address these gaps, we will test a novel 8-week pilot RCT of a non-calorie-restricted whole foods diet adapted from the 2020-2025 Dietary Guidelines for Americans that offers a simple, customizable MyPlate Plan approach (i.e., 5 daily food group goals) focused on individual, family, cultural, and budgetary preferences. We will recruit 30 eligible adolescent (10-18 years) and parent (≥25 years) pairs to test the diet's effects on 1) adolescent body adiposity measured with dual-energy x-ray absorptiometry (DXA) to measure fat mass and anthropometry to measure weight, BMI, and waist circumference (Aim 1) and 2) adolescent and parent diet quality scores measured from dietary recalls using the 2020 Healthy Eating Index during the intervention (Aim 2). Post-intervention family focus groups will be conducted to understand how individual/family needs and preferences and SDOH may be perceived barriers or facilitators of diet adherence in families (Aim 3). Feasibility, acceptability, enrollment, retention, and diet satisfaction data will be generated to establish successful benchmarks to support future studies. Participants randomized to the intervention will receive bi- weekly food delivery, menus, and dietetic support for 8 weeks. Participants randomized to the usual care group will receive a single dietetic counseling session on MyPlate. The successful completion of this study will result in the generation of quantitative and qualitative data to support a future R01 that will test the long-term effectiveness of a whole foods diet on obesity and metabolic outcomes, and diet sustainability in adolescents with obesity and their families.

ELIGIBILITY:
Inclusion Criteria:

For this study, eligible adolescents will be those that:

1. 10-18 years of age at time of initial screening;
2. living at home full-time with the enrolled parent or caregiver (≥80% in primary residence);
3. obesity defined as a body mass index (BMI) greater than or equal to 95th percentile for age and gender based on standardized CDC growth curves;
4. reside within greater Middle Tennessee area and has enrolled parent/caregiver willing to drive to Vanderbilt University and Vanderbilt University Medical Center for study visits;
5. are without medical conditions that would limit participation in a diet-related study (e.g., tube feeding, dysphagia, severe food allergy to 3 or more food groups causing anaphylaxis);
6. are willing and able to participate in an 8-week diet study that encourages preparing and eating healthy foods and snacks for 8 weeks with parental or caregiver support;
7. have parental or caregiver commitment to participate in the research study;

For this study, eligible adult parents or caregivers will be those that:

1. adult parent or primary legal caregiver (greater than or equal to 25 years of age) of an enrolled adolescent;
2. live with the adolescent full-time (≥80% in primary residence);
3. have 1 or more metabolic risk factor(s) and/or metabolic condition(s) (e.g., overweight/obesity, hypertension, hypercholesterolemia or dyslipidemia, hyperglycemia [elevated fasting blood glucose ≥100 mg/dL] and/or prediabetes, history of gestational diabetes, polycystic ovarian syndrome, type 2 diabetes, non-alcoholic fatty liver disease);
4. reside within greater Middle Tennessee area and are willing to drive to Vanderbilt University and Vanderbilt University Medical Center for study visits;
5. are without medical conditions that would limit participation in a diet-related study (e.g., tube feeding, dysphagia, severe food allergy to 3 or more food groups);
6. are able to participate in a study program that encourages preparing and eating healthy foods and snacks for 8 weeks with most preparation/cooking of meals/snacks at home;

Exclusion Criteria:

Adolescent exclusion criteria include:

1. Outside of the specified age range;
2. not living in the home of the enrolled parent or caregiver full time (≥80% in primary residence);
3. BMI less than 95th percentile for age and gender;
4. pregnant or lactating;
5. no eligible enrolled parent or caregiver or lack of parental/caregiver commitment to participate in study;
6. food allergy to 3 or more food groups; dietary restrictions or medical condition that prohibits participation in a diet study;
7. use of medications that cause weight loss or diabetes medications;
8. active participation in a weight loss or intense lifestyle modification program;
9. limited English-language proficiency;
10. participants unwilling or unable to give informed consent, accept random assignment, attend dietary counseling sessions, adhere to treatment prescription, or complete study measures;
11. adolescents who display dissenting behaviors during baseline data collection;
12. adolescents who do not otherwise meet the eligibility criteria listed in sections above as determined by pre-screen;

Adult Parent or Caregiver exclusion criteria include:

1. not parent/ or legal caregiver;
2. not living in a household full-time with enrolled adolescent (less than 80% time spent away from primary residence);
3. lack of metabolic condition(s) per inclusion criteria;
4. special dietary restrictions, food allergies, or medical conditions that prohibit participation in a diet-related study;
5. limited English-language proficiency;
6. participants unwilling or unable to give informed consent, accept random assignment, attend dietary counseling sessions, adhere to treatment prescription, or complete study measures;
7. parent or caregivers who do not otherwise meet the eligibility criteria listed in sections above as determined by pre-screen;

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in adolescent body composition | Baseline to 8-weeks
  Body adiposity will be measured using DXA at the VUIIS with a Hologic Horizon series W scanner (Marlborough, MA). Total body fat mass (primary outcome), trunk fat mass, lean body mass (LBM) in kg, and total body %fat will be recorded.

SECONDARY OUTCOMES:
Changes in adolescent and adult diet quality | Baseline to 8-weeks
  The 2020 Healthy Eating Index (HEI) will be used to estimate adolescent and adult diet quality scores during the study. Scores will be calculated from 3-day food diaries imputed into NDSR software. The HEI uses a scoring system of 0-100 to determine how well an individual's diet (ages ≥2 years) aligns with major DGA recommendations with a higher diet quality score indicating a healthier diet. Dietary information from 3-day food diaries will be used to estimate the baseline diet quality score.
Change in Adult Body Mass Index (BMI) | Baseline to 8-weeks
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. BMI is interpreted using standard weight status categories. These categories are the same for men and women of all body types and ages. Below 18.5 : Underweight; 18.5 - 24.9: Normal or Healthy Weight; 25.0 - 29.9: Overweight; 30.0 and Above: Obese.
Change in adolescent Body Mass Index (BMI) percentiles | Baseline to 8-weeks
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. BMI is interpreted using standard weight status categories. The CDC BMI-for-age charts for children above 2 years will be used to calculate BMI percentiles.
Change in adolescent Body Mass Index (BMI) Z Scores | Baseline to 8-weeks
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. BMI is interpreted using standard weight status categories. The CDC BMI-for-age charts for children above 2 years will be used to calculate BMI z-scores.
Change in adolescent and adult Waist Measurements | Baseline to 8-weeks
  Waist circumference will be measured in centimeters.
Diet adherence in adolescents and adults | Baseline to 8-weeks
  ≥80% compliance with the diet will be considered "adherent" and will be estimated qualitatively from food diaries. The dietitian will review food checklists/diaries to assess adherence and to modify diets or support compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Sneed, PhD, MSN, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University School of Nursing, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No